| Structural Types of the Foot and Their Influence on Core and Sports Performance in College Athletes |
|---|
| NCT ID not yet assigned |
| Date: 25/August/2022 |

## **INFORMED CONSENT**

Researchers' Names: Orlando Santiago Moreno Barriga Date: 08/10/2022

Research Title: Characterization of the Medical-Sports Condition Variables, Physical Performance, and Neuromuscular Response of Representative Athletes from the University of Magdalena

Research Objective: To understand the basic medical, physical condition, and sports performance of representative student athletes from the University of Magdalena in order to characterize their current physical and medical condition.

Instruments to be Used to Obtain Results: A complete medical-sports history will be taken using basic medical equipment from the Sports Medicine office, including anthropometric measurement devices. Additionally, non-invasive measurement equipment for motion analysis and functional evaluation of posture, stability, and balance will be used. Timing equipment will measure race times and speed, and equipment will be used to measure neuromuscular activity, strength, and joint function, as well as the athletes' aerobic performance.

Benefits of Participating in the Research: By understanding the medical and physical condition of the athletes, programs and protocols can be developed to improve their physical condition, health, and contribute to enhancements in sports performance.

Possible Risks of Participating: The risks are inherent to the performance of physical exertion tests and conducting physical work similar to what is done in the field.

Access to Information: Only the researchers have access to the information.

Who Will Know the Results: The results of this research will be known by the researchers and the sports community, as well as coaching staff. Additionally, since this study is part of research, it is intended to be shared with the interested community through possible publication in a scientific journal, without disclosing the names of the participants in the study.

| Who Can I Contact if I Have Any Questions: You car | directly contact the researchers Orlando Moreno. |
|---|---|
| I, | · |
| Participant's Signature | |